CLINICAL TRIAL: NCT07316764
Title: Eccentric Cycling : a New Training Modality in Multiple Sclerosis Rehabilitation
Brief Title: Eccentric Cycling in Multiple Sclerosis Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: University Hospital Sart Tilman, Liege (Unknown)
Responsible Party: Principal Investigator, Vandenbroeck Benoit, Physiotherapist, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-416
Record Dates: First submitted 2025-12-08; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Rehabilitation; Neuro-Degenerative Disease; Neurorehabilitation
Keywords: eccentric cycling; multiple sclerosis; eccentric training; neurorehabilitation; physical therapy; neuro-degenerative disease
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Participants will be split in 2 groups :
  one following an eccentric cycling training one following a concentric cycling training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric group (Experimental)
  Interventions: Other: Eccentric training
- Concentric group (Active Comparator)
  Interventions: Other: Concentric training

INTERVENTIONS:
Other: Eccentric training — Eccentric cycling training
  Arms: Eccentric group
Other: Concentric training — Concentric cycling training
  Arms: Concentric group

SUMMARY:
The project aims to optimise functional rehabilitation programmes for people with multiple sclerosis.

Investigators are proposing eccentric cycling as a new exercise modality for treating these patients.

Based on previous results in healthy subjects, investigators will attempt to define the optimal parameters of this new modality (in terms of duration, intensity, frequency, etc.).

Investigators also aim to demonstrate the effectiveness of this training (compared to conventional training) in improving muscle function, functional capacity, perception of chronic fatigue, quality of life, physical condition, and neurological and cognitive function.

DETAILED DESCRIPTION:
Our study will focus on multiple sclerosis. For each pathology included, a "control" group will consist of patients undergoing a traditional rehabilitation program combined with a concentric cycling session. An experimental group ("eccentric rehabilitation") will consist of patients enrolled in an eccentric ergocycle training protocol paired with standard rehabilitation. In practice, a portion of the classical rehabilitation program will be replaced by either concentric or eccentric cycling, for a maximum duration of 30 minutes. Based on a preliminary study conducted in healthy subjects, a review of the existing literature, and a sample size calculation performed by the Biostatistics Department of the University Hospital of Liège, investigators aim to recruit 60 to 80 subjects per pathology (details in the appendix). Participation of pregnant women is permitted.

Type of Study

This is a prospective interventional study conducted longitudinally, with all subjects evaluated over the same time period (2025-2027). The study will take place at the Sart-Tilman sites (Blanc-Gravier, Exercise Physiology Unit) or at the CNRF in Fraiture-en-Condroz, depending on participant preference.

Neurological Pathologies Inclusion criteria

Participants must:

present with one of the following neurological disorders: Parkinson's disease or multiple sclerosis.

I. Eccentric Rehabilitation Program

Given the increasing clinical interest in eccentric contraction modalities for chronic diseases, a semi-recumbent eccentric ergometer has been specifically designed for clinical use. Patient installation on this device is safe and easily achievable, and the semi-recumbent position provides additional comfort during exercise. The ergometer allows secure workload control via visual feedback powered by dedicated software. The device can be transported between sites (Sart-Tilman - Fraiture - Esneux).

Experimental Protocol

This experimental study aims to establish and compare the effects of an eccentric cycling training protocol versus a traditional concentric cycling protocol performed on an ergometric bicycle. Subjects will be randomly allocated (stratified by sex and disease stage) into one of the two experimental groups. Randomization will be conducted by Mr. Benoît Vandenbroeck after encoding the relevant data in a table and assigning subjects within each stratum using random distribution.

Participants will undergo a 2-week evaluation period followed by a 12-week training program consisting of two sessions per week, for a total of 28 sessions. Sessions will take place either at the Neurological and Functional Rehabilitation Center in Fraiture-en-Condroz (CNRF) or at Blanc-Gravier (Sart-Tilman), according to participant preference. Training sessions (eccentric or concentric) will last a maximum of 30 minutes. For participants already enrolled in a rehabilitation program at the CNRF, part of their traditional session will be replaced by the cycling training.

The unusual nature of eccentric training may induce mild delayed-onset muscle soreness (DOMS), including pain and stiffness, appearing 24-48 hours after exercise. These symptoms are transient, and symptomatic treatments (analgesics, stretching, ice) are not permitted.

Multiple variables will be assessed before, during, and after the intervention period to quantify potential effects of each training protocol and allow direct comparison.

Description of Study Phases

The study consists of 5 phases over a 12-week period (see appendix):

Phase 0: Baseline Testing

Measurements will be collected 5-7 days before and 7-14 days after the training period to monitor longitudinal changes and evaluate the impact of the protocols on body composition and functional capacity.

Eccentric Ergocycle Training Protocol Phase 1: Familiarization (4 weeks)

Two sessions per week for four weeks. The main objective is to familiarize subjects with eccentric cycling and its specific neuromuscular demands, thus limiting potential muscle damage. Duration and intensity will gradually increase. To progress to the training phase, subjects must maintain an average power output within ±10% of their target theoretical power during the final familiarization session. If needed, one to two additional weeks of familiarization may be added. Beyond this point, participants unable to meet the criteria will be withdrawn from the study.

Phase 2: Training (Part 1 - 4 weeks)

These four weeks establish the first phase of training, with predefined duration and intensity levels.

Phase 3: Training (Part 2 - 4 weeks)

An additional four weeks are included, based on evidence showing greater benefits after 8-12 weeks of training. Intensity will be increased during this phase.

Throughout the 12-week training period, temporal progression and identification of potential physiological adaptations will be monitored.

Phase 4: Final Testing

Participants will return to the laboratory twice to repeat the baseline assessments. These tests will be performed 7-10 days after the final training session to ensure adequate muscle recovery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* Multiple sclerosis: EDSS score < 7
* Age under 75 years
* Stable disease state
* Written medical clearance authorizing participation
* Legal adult status
* Written informed consent, with demonstrated understanding of the consent form (via a few specific questions)
* Ability to mobilize independently (e.g., transfers, walking)

Exclusion Criteria:

* One or more contraindications to physical activity
* Significant comorbidities
* Current hospitalization or undergoing changes in medication
* Active flare-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximal Isometric Force | At baseline and endline of intervention (Week 1 and 14)
  Maximal Isometric Force (in Newton-meters - Nm) of the quadriceps will be measured using a fixed dynamometer (Kinvent), at 90 degrees of knee flexion.
Walking distance | At baseline and endline of intervention (Week 1 and 14)
  6 minutes walking test and 2 minutes walking test will be performed to measure the walking capacities (in meters) of participants.

SECONDARY OUTCOMES:
Handgrip strength | At baseline and endline of intervention (Week 1 and 14)
  Handgrip strength (in kilograms) will be measured using a handheld dynamometer.
Spasticity | At baseline and endline of intervention (Week 1 and 14)
  Spasticity will be evaluated using the Tardieu's scale of spasticity (expressed in arbitrary unit).
  This scale ranges from 0 (no resistance) to 4 (immobile)
Timed up and go | At baseline and endline of intervention (Week 1 and 14)
  The TUAG (in seconds) will be used to evaluate lower limb functional capacity
Neurocognitive capacity | At baseline and endline of intervention (Week 1 and 14)
  Neurocognitive capacity will be evaluated using a combinaison of Tests of Attentional Performance battery (TAP battery)
Berg Balance Scale | At baseline and endline of intervention (Week 1 and 14)
  The balance test will be used to evaluate balance capacity (expressed in arbitrary unit). This scale ranges from 0 (High fall risk) to 56 (no fall risk)
Five time sit to stand test | At baseline and endline of intervention (Week 1 and 14)
  The sit to stand test (in seconds) will be performed to measure lower limb functional capacity
Maximal aerobic power | At baseline and endline of intervention (Week 1 and 14)
  Maximal aerobic power (in Watts) will be evaluated by performing a Cardiopulmonary Exercise Test on an ergocycle.
Maximal oxygen consumption | At baseline and endline of intervention (Week 1 and 14)
  Oxygen consumption (in milliliter per minute per kilogram ) will be evaluated by performing a cardiopulmonary exercise test on an ergometer.
Fatigue | At baseline and endline of intervention (Week 1 and 14)
  Fatigue will be evaluated using the modified fatigue impact scale (MFIS) (expressed in arbitrary unit). This scale present different item that should be ranged from 0 (never) to 4 (always). We will collect the physical aspect with a maximal score ranginig from 0 (no fatigue) to 36 (exhausted)
Multiple Sclerosis Quality of Life-54 | At baseline and endline of intervention (Week 1 and 14)
  Quality of life will be evaluated using the Multiple Sclerosis Quality of Life-54 (MSQoL-54). This scale will be expressed in percent.
Maximal heart rate | At baseline and endline of intervention (Week 1 and 14)
  Maximal heart brate (in beats per minute) will be measured by performing a cardiopulmonary exercise test on an ergocycle.

OTHER OUTCOMES:
Height | At baseline and endline of intervention (Week 1 and 14)
  Height will me measured and expressed in centimeters.
Weight | At baseline and endline of intervention (Week 1 and 14)
  Weight in kilograms will be measured using a Tanita scale.
Body fat percentage | At baseline and endline of intervention (Week 1 and 14)
  Body fat percentage (in percent) will be measured using a Tanita scale.
Body mass index | At baseline and endline of intervention (Week 1 and 14)
  BMI (in kilograms per square meters) will be measured using the height and the weight (H/W^2).
Heart rate | Throughout the entire intervention (week 2 to week 13)
  Heart rate (in percent of max heart rate) will be analyzed during each training session
Rating of perceived exertion | Throughout the entire intervention (week 2 to week 13)
  RPE (in arbitrary unit) will be evaluated using the Borg scale after each training session. Borg scale ranges from 6 (no exertion) to 20 (extremely hard).
Mental demand | Throughout the entire intervention (week 2 to week 13)
  Mental demand of the training (in arbitrari unit) will be evaluated using a modified Borg scale after each training session. Modified Borg scale ranges from 0 (no exertion) to 10 (extremely hard).
Muscle soreness | Throughout the entire intervention (week 2 to week 13)
  Muscle soreness (in arbitrary unit) will be evaluated using a visual analog scale before each training session. This scale ranges from 0 (no pain) to 10 (worst pain possible).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie HODY, PhD, Study Chair — Department of Physical Activity and Rehabilitation Sciences, University of Liege and University Hospital of Liege, Liege, Belgium
Locations (1):
- Liege University, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No